CLINICAL TRIAL: NCT01413867
Title: Safety and Short Term Effectiveness of EEA Stapler vs PPH Stapler in the Treatment of III Degree Haemorrhoids. Prospective Randomized Controlled Trial
Brief Title: Safety and Short Term Effectiveness of EEA Versus PPH Stapler for III Degree Hemorrhoids
Acronym: EEA/PPH2011
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Societa Italiana di Chirurgia ColoRettale (Network)
Responsible Party: Principal Investigator, Donato F Altomare, Associate professor, Societa Italiana di Chirurgia ColoRettale
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: No sponsor
Record Dates: First submitted 2011-08-08; First posted 2011-08-10 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: III Degree Hemorrhoids
Keywords: hemorrhoids; circular staplers; mucosal resection; hemostatic suture
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- EEA group (Experimental): Group of patients with III degree hemorrhoids treated by EEA stapler
  Interventions: Procedure: stapled hemorrhoidopexy
- PPH group (Active Comparator): group of patients with III degree hemorrhoids treated by PPH stapler
  Interventions: Procedure: stapled hemorrhoidopexy

INTERVENTIONS:
Procedure: stapled hemorrhoidopexy — stapled hemorrhoidopexy will be performed using the EEA stapler Covidien
  Arms: EEA group
Procedure: stapled hemorrhoidopexy — stapled hemorrhoidopexy will be performed using the PPH01/03 Ethicon EndoSurgery
  Arms: PPH group

SUMMARY:
Stapled hemorrhoidopexy has gained wide acceptability among colorectal surgeons because of less postoperative pain compared with excisional surgery, however a still relevant percentage of postoperative bleedings and long-term hemorrhoid recurrence are reported. A new stapler device has been designed to overcome these drawbacks by modifying the stapled sutures and by increasing the space for mucosal resection in the case of the stapler.

This randomized controlled study was aimed to demonstrate whether the new EEA stapler Covidien was able to resect more quantity of prolapsed mucosa than the traditional PPH 01/03 Ethicol Endosurgery by measuring the surface of the resected specimen and to demonstrate if the modified stapled sutures can ensure better intraoperative hemostasis by measuring the number of overstitches required to get perfect hemostasis during the operation.

ELIGIBILITY:
Inclusion Criteria:

* III degree Hemorrhoids
* written informed consent
* mental ability to understand the procedure

Exclusion Criteria:

* Previous treatments for hemorrhoids or other proctological diseases
* Fecal Incontinence
* Chronic inflammatory bowel disease
* Anal sphincter lesions
* coagulative defects
* obstructed defecation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
quantity of anorectal mucosa resected using two different circular staplers | 1 hour following the end of the operation
  The surface (in cm2)of anorectal mucosa resected during stapled hemorrhoidopexy for III degree hemorrhoids, using two different circular staplers will be compared

SECONDARY OUTCOMES:
Number of hemostatic stitches required to get perfect hemostasis using 2 different staplers | 1 hour after each operation
  the number of hemostatic sutures required to get perfect hemostasis during stapled hemorrhoidopexy using 2 different staplers for III degree hemorrhoids

CONTACTS AND LOCATIONS:
Locations (1):
- Dept of Emergency and Organ transplantation, Bari, Italy